CLINICAL TRIAL: NCT02333279
Title: Cancer Development In Organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other); Cantonal Hospital of St. Gallen (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: FUP062; snctp000000587 (Other: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2014-12-18; First posted 2015-01-07 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Heart Cancer; Kidney Cancer; Lung Cancer; Pancreas Cancer; Liver Cancer
MeSH Terms: conditions — Heart Neoplasms; Kidney Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Organ transplant recipients: Follow-ups in regular intervals following the organ transplant date.

SUMMARY:
The investigators will determine the cancer risk in organ transplant recipients compared to the general population with the help of statistical analysis. Secondly the investigators will try to characterize the different cancer types.

DETAILED DESCRIPTION:
This cohort analyses will focus on incident and recurrent cases of development of non-skin cancer over time. We will consider time to first formation of non-skin solid cancer after solid organ transplantation as well as the cumulative number of non-skin solid cancer formation over time. Both aspects are equally important and will be reflected in the analytic methods of this study. Theses analyses will be restricted to the most prevalent transplantation types of heart, kidney, liver, and lung.

ELIGIBILITY:
Inclusion Criteria:

We will select all patients within the STCS based on the date of the first solid organ transplantation. Patients with multiple organ transplantations will be included as well. Patients contribute to the study observation time until death or end of follow-up due to other reasons.

Exclusion Criteria:

We will exclude patients with non-solid organ transplantation (e.g. hematopoietic stem cell transplantation), because the detailing of information in the STCS is insufficient to allow for detailed analysis of cancer development and control of relevant confounders. We will exclude

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All solid organ transplant recipients in Switzerland since 2008 who have given their consent to be included in the study.
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Number of solid cancers | Ten Year followup
  Number of solid cancers

CONTACTS AND LOCATIONS:
Overall Officials: Gunther FL Hofbauer, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Switzerland

REFERENCES:
- [Result] Lengwiler E, Stampf S, Zippelius A, Salati E, Zaman K, Schafer N, Schardt J, Siano M, Hofbauer G, The Swiss Transplant Cohort Study. Solid cancer development in solid organ transplant recipients within the Swiss Transplant Cohort Study. Swiss Med Wkly. 2019 May 19;149:w20078. doi: 10.4414/smw.2019.20078. eCollection 2019 May 6. PMID 31104307